CLINICAL TRIAL: NCT00223834
Title: Pathways to Vocational Rehabilitation: Enhancing Entry and Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Drebing, Charles - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E3436R
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Poverty; Unemployment
Keywords: Counseling; Motivation; Psychotherapy, brief

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Single session orientation to available services
  Interventions: Behavioral: single session of Motivational Interviewing

INTERVENTIONS:
Behavioral: single session of Motivational Interviewing

SUMMARY:
This study will examine the barriers and supports for entering and receiving work-related services for veterans with a serious mental illness. It will also determine the effectiveness of a brief motivational interviewing intervention designed to help veterans receive these services.

DETAILED DESCRIPTION:
Randomized clinical trials and naturalistic studies show that among patients meeting criteria for chronic mental illness, those participating in vocational rehabilitation (VR) have significantly reduced days of inpatient hospitalization. Unfortunately, the majority of eligible adults fail to enter VR and almost half of those who do, drop out or are involuntarily discharged. The reasons for nonparticipation and drop out and their impact on rehabilitation outcomes are poorly understood.

The study will provide needed naturalistic data documenting:

1. the way in which barriers function to reduce entry to services and contribute to the high rate of dropout,
2. the outcomes associated with different patterns of participation, and
3. relative rates of entry and retention in a non-VHA VR exemplar of the Intensive Placement and Support (IPS) model at the Manchester Mental Health Center in Manchester, New Hampshire.

While we need to know more about these "barriers" in order to develop the range of appropriate interventions, the enhancement of client motivation for work and rehabilitation is likely to have a positive impact both on entry and sustained compliance. We are proposing a random assignment single blind trial of a brief Motivational Interviewing (MI) intervention designed to address the low entry and retention rates of veterans with Serious Mental Illness (SMI) in Veterans Health Administration's (VHA) VR services.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of serious mental illness, present for at least 2 years
* Is unemployed or underemployed
* Current episode of un/underemployment is at least 3 months
* Enrolled to receive services at study site

Exclusion Criteria:

* Over the age of 55
* Non-English speaker
* Mini-Mental score of less than 20
* Planning to move more than 30 miles from study site in the next 18 months
* Previously screened for this study
* Currently or previously involved in other research studies which may impact variables relevant to this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Entry and Retention in Vocational Rehabilitation | 18 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charles Drebing, PhD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Bedford, Massachusetts, United States